CLINICAL TRIAL: NCT01541943
Title: A Phase 3, Randomized, Double- Blind, Multi-center, Double Dummy, Clinical Trial Comparing HL-040XC With Single Component Therapies(Atorvastatin, Losartan) to Assess the Efficacy and Safety of HL-040XC in Patients With Essential Hypertension and Hyperlipidemia
Brief Title: Efficacy and Safety of HL-040XC in Essential Hypertension and Hyperlipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HanAll BioPharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HATLO11III_1
Record Dates: First submitted 2012-02-24; First posted 2012-03-01 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Essential Hypertension; Hyperlipidemia
Keywords: Atorvastatin; Losartan; Essential Hypertension; Hyperlipidemia
MeSH Terms: conditions — Essential Hypertension; Hyperlipidemias | interventions — Atorvastatin; Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- HL-040XC (Experimental): Once daily, administered orally, 8 week
  Interventions: Drug: HL-040XC
- Atorvastatin (Active Comparator): Once daily, administered orally, 8 week
  Interventions: Drug: Atorvastatin
- Losartan (Active Comparator): Once daily, administered orally, 8 week
  Interventions: Drug: Losartan
- Placebo (Placebo Comparator): Once daily, administered orally, 8 week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Once daily, administered orally, 8 week
  Other Names: Lipitor
  Arms: Atorvastatin
Drug: Losartan — Once daily, administered orally, 8 week
  Other Names: Cozaar
  Arms: Losartan
Drug: Placebo — Once daily, administered orally, 8 week
  Arms: Placebo
Drug: HL-040XC — Once daily, administered orally, 8 week
  Arms: HL-040XC

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of HL-040XC in patients with essential hypertension and hyperlipidemia

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 80 years
* History of essential hypertension and hyperlipidemia
* Able to sign informed consent

Exclusion Criteria:

* At screening, SBP ≥ 180mmHg or DBP ≥ 110mmHg or LDL-C > 250mg/dL or TG ≥ 400mg/dL
* Has a history of hypersensitivity to Angiotensin Ⅱ receptor blocker or HMG-CoA reductase inhibitor or component of this drug

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2012-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline to 8 week in SiDBP (Sitting Diastolic Blood Pressure) | Baseline and 8 week
Percent change from baseline to 8 week in LDL-Cholesterol | Baseline and 8 week

SECONDARY OUTCOMES:
Percentage of patients reaching treatment goals according to NCEP ATP III Guideline and Blood Pressure Responder according to JNC VII Guideline. | Baseline and 4, 8 week

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Gyu Park, Medicine, Principal Investigator — Department of Cardiovascular, Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, Seoul, South Korea